CLINICAL TRIAL: NCT04789057
Title: Non-commercial Clinical Trial of Statins CAncer Preventive and Pleiotropic TherApy IN Smokers With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Atorvastatin Effect on Reduction of COPD Exacerbations
Acronym: Captain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/ABM/01/00074; 2019/ABM/01/00074 (Other: Medical Research Agency)
Record Dates: First submitted 2021-02-15; First posted 2021-03-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Copd; COPD Exacerbation; Smoking; Gene Expression; Atorvastatin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statins (Experimental): Atorvastatin 40 mg treatment, p.o., QD
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Placebo (Placebo Comparator): Placebo tablet, p.o., QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — p.o., once daily
  Other Names: Atorvastatin
  Arms: Statins
Drug: Placebo — p.o., once daily
  Other Names: Placebo control group
  Arms: Placebo

SUMMARY:
It is a randomized, multicenter, prospective, double-blind, placebo controlled, interventional clinical trial that will be conducted in Poland, in about 12 Hospital Pulmonary Departments to evaluate the effectiveness of atorvastatin on the reduction of inflammation process in patients with chronic obstructive pulmonary diseases, and possible biomarkers for personalized treatment of COPD.

DETAILED DESCRIPTION:
It will be a randomized, double-blind, two arm clinical study to assess effect of atorvastatin 40 mg treatment in patients with stable COPD. The whole study duration will include three phases: pre-study screening and enrollment procedures (4 weeks), clinical assessment at dosing (52 weeks), and post study follow up (4 weeks). During the participation in the study subjects will attend Visit 1 (V1, -4 weeks), visit 2 (V2, day 0), visit 3 (V3, week6), visit 4 (V4, week 12), visit 5 (V5, week 26), visit 6 (V6, week 38), visit 7 (V7, week 52), and follow-up end of study visit (EOS, 56 weeks). The study will begin with a 4-weeks screening phase where patients who fulfill preliminary inclusion/exclusion criteria (prior to entry into study), will be given informed consent and screened. The baseline laboratory tests, clinical and medical evaluation including concomitant medication and drug of abuse will be completed to determine patient continuing eligibility to participate in the study.

Upon confirmation of eligibility, the patients will be randomized into two treatment groups receiving one of two medications tested in the study. Each patient enrolled into the clinical study will have to report to the clinic 7 times in order to complete procedures. Blood will be drawn before and during the statin or placebo treatment from patients according to study protocol. This part of the project aims to develop statin response biomarkers for personalized treatment of COPD, based on RNA-sequencing (RNA-seq) information derived from, leukocytes and blood plasma of COPD patients with characterized clinical Atorvastatin response phenotypes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed Informed Consent Form and is able to understand the purpose and procedures required for the study and is willing to participate in the study.
2. Subject [male or female] is aged 40 years and older.
3. Subject is able to understand and comply with the protocol requirements and instructions and is likely to complete the study as planned.
4. Patients with stable COPD with persistent airflow limitation (stable COPD (post-bronchodilator FEV1<80% of the predicted normal and post-bronchodilator FEV1/FVC<0,70 at visit 1.) Stage II- IV) and with moderate to very severe airflow limitation according to GOLD guidelines.
5. At least two moderate/severe COPD exacerbations, or at least one leading to hospitalization or ICU admission within 12 months, preceding screening visit.
6. Current or ex-smokers who have a smoking history of at least 10 pack years.

Exclusion Criteria:

1. Contraindication to statin therapy included but not limited to: known poliomyelitis, motor neuron disease, cranial or temporal arteritis, stroke or myopathy.
2. Statin use within the last 3 months prior to study start.
3. Prior diagnosis of statin induced myopathy or hypersensitivity reaction to another HMG-CoA-reductase inhibitor.
4. Using e-cigarettes or I IQOS tobacco heating system.
5. Pregnant or nursing (lactating) women.
6. Women of child bearing potential, unless they are using effective method of contraception during dosing of study treatment.
7. Patient with a clinically significant abnormality at visit 1 in investigator opinion.
8. Patients with a clinically relevant laboratory abnormality at visit 1 in investigator opinion.
9. Patients with a history of malignancy of any organ system (including lung cancer).
10. Patients unable to perform acceptable spirometry and lung volumes procedures.
11. Patients who had a COPD exacerbations that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the 6 weeks prior to visit 1.
12. Patients who have had a respiratory tract infection within 4 weeks prior to visit1.
13. Patients requiring oxygen therapy (>15hr/day) on a daily basis for chronic hypoxemia.
14. Patients with a history of asthma or onset of symptoms prior to age 40 years
15. Patients with concomitant pulmonary disease (e.g. lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, tuberculosis).
16. Patients with primary bronchiectasis.
17. Patients with a diagnosis of α-1 antitrypsin deficiency (AATD).
18. Patients with pulmonary lobectomy or lung volume reduction surgery or lung transplantation.
19. Active abuse of drugs or alcohol, poor compliance anticipated.
20. Use concomitant medications that are known to interact with atorvastatin: warfarin and other coumarin (vitamin K antagonists) anticoagulants, cyclosporin, gemfibrozil or other non or selective nonsteroidal anti-inflammatory drugs, proton pump inhibitors (PPIs) used by last 6 months.
21. Patients participating in or planning to participate in the active phase of a supervised pulmonary rehabilitation program during the study.
22. Use of other investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening visit.
23. Those unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbation rate | 56 weeks
  The exacerbation of the disease (defined as an acute worsening of respiratory symptoms that results in additional therapy) will be measured during the study treatment and follow-up phases, and compared between studied groups.
Time to the COPD exacerbation | 56 weeks
  The time to the first exacerbation will be compared between the Intervention and Placebo groups.

SECONDARY OUTCOMES:
Changes in forced expiratory volume in the first second (FEV1) | 56 weeks
  The differences in absolute value between Placebo and Atorvastatin group will be evaluated in time points [Visit 1 ,Visit 3,Visit 4, Visit 5, Visit 6 and Visit 8], and the relative change between Visit 1 and following time points [Visit 3 - Visit 8] in both arms will be compared.
Changes in health-related quality of life | 56 weeks
  The St George's Respiratory Questionnaire (SGRQ) score will be used and the differences in absolute value between Placebo and Atorvastatin group will be evaluated in time points [Visit 2 , Visit 5, and Visit 7], as well as the - relative change between Visit 2 and following time points [Visit 5 and Visit 7] in both arms will be compared. Scores range from 0 to 100; higher scores indicating more limitations.
Changes of inflammatory pathway gene expression | 56 weeks
  The gene expression will be evaluated in the peripheral blood leucocytes (PBL) by RNA-seq analysis, at visit Visit 1, Visit 2, Visit 5 and Visit 7, and the differences between Placebo and Atorvastatin groups will be analyzed, as well as a relative change between visits Visit 1 and Visit 2, Visit 5 and Visit 7 in both arms will be compared.
Changes in peripheral blood leucocyte count | 56 weeks
  The peripheral blood leucocytes count will be measured and the differences in absolute values between Placebo and Atorvastatin group will be calculated in time points Visit 1 ,Visit 3, Visit 5 and Visit 7, as well as a relative change between visits Visit 1 and Visit 2, Visit 3, Visit 5 , Visit 7 in both arms will be compared.
Changes in the blood fibrinogen concentrations | 56 weeks
  A blood fibrinogen concentration will be measured and the differences in absolute values between Placebo and Atorvastatin group will be calculated in time points Visit 1 ,Visit 3, Visit 5 and Visit 7, as well as a relative change between visits Visit 1 and Visit 2, Visit 3, Visit 5 , Visit 7 in both arms will be compared.
Changes in the blood Interleukin-6 concentrations | 56 weeks
  The Interleukin-6 blood concentrations will be measured and the differences in absolute values between Placebo and Atorvastatin group will be calculated in time points Visit 1 ,Visit 3, Visit 5 and Visit 7, as well as a relative change between visits Visit 1 and Visit 2, Visit 3, Visit 5 , Visit 7 in both arms will be compared.
Changes in the blood high sensitivity C - reactive protein concentrations | 56 weeks
  The blood high sensitivity C - reactive protein concentrations will be measured and the differences in absolute values between Placebo and Atorvastatin group will be calculated in time points Visit 1 ,Visit 3, Visit 5 and Visit 7, as well as a relative change between visits Visit 1 and Visit 2, Visit 3, Visit 5 , Visit 7 in both arms will be compared.

OTHER OUTCOMES:
Change from baseline in pre-dose values of plethysmography | 56 weeks
  The functional residual volume (FRC) will be evaluated at Visit 2, Visit 5 and Visit 7, and changes from Visit 1 will be calculated, as well as compared between studied groups.
Change in Inspiratory capacity (IC) | 56 weeks
  The Inspiratory capacity (IC) will be evaluated will be evaluated at Visit 2, Visit 5 and Visit 7, and changes from Visit 1 will be calculated, as well as compared between studied groups.
Change in 6 minute walking distance (6MWD) test result | 56 weeks
  The 6MWD tests will be performed at Visit 2, Visit 5 and Visit 7, and changes from Visit 1 will be calculated, as well as compared between studied groups.
The rate of hospitalizations (pulmonary or MACE) | 56 weeks
  The number of hospitalizations during the treatment and follow-up phases will be evaluated, and compared between studied groups.
Changes in blood pressure | 56 weeks
  The changes in blood pressure from Visit 1 will be evaluated at Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7, and changes from Visit 1 will be calculated, as well as compared between studied groups.
Changes in heart rate (HR) | 56 weeks
  The changes in HR from Visit 1 will be evaluated at Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7, and changes from Visit 1 will be calculated, as well as compared between studied groups.
Changes in hematology results | 56 weeks
  The changes in hematology results from visit Visit 1 will be evaluated, at Visit 3, Visit 5, and Visit 7, as well as the differences between studied groups will be compared.
Changes in biochemistry results | 56 weeks
  The changes in biochemistry results from visit Visit 1 will be evaluated, at Visit 3, Visit 5, and Visit 7, as well as the differences between studied groups will be compared.
Changes in lipids profile | 56 weeks
  The changes in lipids profile results from visit Visit 1 will be evaluated, at Visit 3, Visit 5, and Visit 7, as well as the differences between studied groups will be compared.
Changes in blood glucose levels | 56 weeks
  The changes in blood glucose concentrations from Visit 1 will be evaluated at Visit 7, and compared between studied groups.
Changes in HbA1c levels | 56 weeks
  The changes in HbA1c levels from Visit 1 will be evaluated at Visit 7, and compared between studied groups.
Changes in the blood AspAT and ALAT concentrations | 56 weeks
  The changes in blood AspAT and ALAT concentrations from Visit 1 will be evaluated, at Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7, and compared between studied groups.
Changes in the blood CPK concentrations | 56 weeks
  The changes in blood CPK concentrations from Visit 1 will be evaluated, at Visit 2, Visit 3, Visit 4, Visit 5, Visit 6 and Visit 7, and compared between studied groups.
Change in a transfer factor of the lung for carbon monoxide (DLCO) | 56 weeks
  The DLCO will be evaluated at Visit 2, Visit 5 and Visit 7, and the changes from Visit 1 will be calculated, as well as compared between studied groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mróz, Prof. MD, Principal Investigator — Medical University of Bialystok
Locations (1):
- Medical University Hospital, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No
According to the agreement with the funding institution (Medical Research Agency), the sponsor and research centers must obtain the consent of the funding institution to disclose the clinical trial data.